CLINICAL TRIAL: NCT04085302
Title: Mixed Methods (Quantitative, Qualitative) Feasability Study Assessing Engagement With the First Version of the TARA Working Prototype (a Digital Behaviour Change Intervention, DBCI) in Individuals With COPD
Brief Title: TARA Working Prototype Engagement Evaluation: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0352-2133
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Device: Digital Behaviour Change Intervention

INTERVENTIONS:
Device: Digital Behaviour Change Intervention — 14 days

SUMMARY:
TARA is a Digital Behaviour Change Intervention (DBCI) for individuals with Chronic Obstructive Pulmonary Disease (COPD)(IwCOPD), which has been designed using a Human-Centred Design (HCD) methodology. HCD involves, among other elements, members of the target audience in evaluations at multiple stages within the design process.

This feasibility study is primarily designed to assess the acceptability of the DBCI test asset to the target audience. Acceptability as defined for the purpose of this study includes usability of the system, and perceived value and desirability to the end-user audience. As such, engagement in this context is deemed to mean the degree to which the test asset provides a usable, acceptable, desirable and valuable experience to its users during a time-limited trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written electronic informed consent (e-consent) in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the study
* Male or female patients
* All patients must have a self-reported confirmation of a physician diagnosis of Chronic Obstructive Pulmonary Disease (COPD)(or chronic bronchitis or emphysema)
* Age ≥ 40 years
* Patients must be current or ex-smokers with a smoking history of at least 10 pack-years (pack years = [cigarettes per day/20] x years of smoking)
* Modified Medical Research Council (mMRC) Score ≥ 1 (i.e. evidence of activity-related breathlessness)
* Patients must have a current prescription for once daily maintenance bronchodilator in keeping with their approved labels as well as a short-acting bronchodilator ("rescue medication") for at least 3 months prior to study enrolment
* Participants must be willing to use a smart watch and be willing to complete all data collection requirements (within TARA plus phone interview plus on-line questionnaires)
* Patients must confirm that his/her treating physician has been informed about the patient's participation in the study (prior to TARA log-in)
* Fluency in written English
* Currently residing in US (for duration of study)
* Not fully adherent (self-report) to once daily inhaled COPD medication (<80% on a protocol-specific participant self-assessment scale of medication adherence (0 - 100%))
* Access to (and comfort with) a digital device (Desktop; Laptop; Tablet), with updated Firefox [version 67.0 and above] or Chrome [version 75.0.3770.80 and above] browsers installed (or willing to download up-to-date version for the study), and daily home access to internet
* Need to have personal e-mail account that is used daily

Exclusion Criteria:

* Patients with asthma
* Patients who are currently prescribed oxygen therapy
* Patients who have completed a pulmonary rehabilitation (PR) program in the 6 weeks prior to enrolment or patients who are currently in a PR program (rationale: PR programs typically include a self-management component which may interfere with study objectives)
* Planned vacation period during the study period that requires overnight stays away from home
* Major surgery performed within 6 weeks prior to enrolment or planned within 2 months after enrolment, e.g. hip replacement
* Previous enrolment in this study
* Currently enrolled in another investigational device or drug study/trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Current use of a Smartwatch and/or wrist-worn step counter and not willing to switch to the study-specific Smartwatch for the duration of study
* Any medical or neuro-cognitive condition that would limit the ability of the participant to consent
* Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
% of study participants achieving 80% or higher engagement score with their personal TARA program | Up to 14 days
Study participant's motivation to engage with the TARA working prototype (version 1) and their perceptions of value and usefulness | Up to 14 days
  Qualitative assessment of motivation and perceptions of value and usefulness at different stages in the participant's journey through the prototype; data sourced via discussion in an exit interview at the end of the study.
Evidence of usability issues, patterns of dis-engagement or failures of use in particular pages or functional areas of the prototype | Up to 14 days
  Analysis of usage data of the site to explore if there are common points at which participants fail to progress, make mistakes or abandon interactions; Data will be sourced from individual and amalgamated usage analytics - data points will include drop-out rates for each of the main functional areas of the site and will be supplemented by within-page usage data An overall score for perceived ease-of-use will be generated using the 'System Usability Scale' (SUS), using self-reported data from the pre- and post-TARA participant questionnaire
Study participant's reports of usability or other issues from using the prototype | Up to 14 days

SECONDARY OUTCOMES:
% of study participants who achieve a score of 8 or greater in Knowledge, Motivation, Confidence (KMC) assessments | Up to 14 days
% of study participants who achieve a positive change in measures of motivation, activation, competence (self-efficacy) and stage of change | Up to 14 days
% of study participants who report increases in adherence to once daily inhaled medication and reduction in Chronic Obstructive Pulmonary Disease (COPD) symptoms | Up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medullan, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/